CLINICAL TRIAL: NCT06938776
Title: Effect of a Musical Toy on Pain, Fear, and Parental Satisfaction During IV Cannulation in Hospitalized Children
Brief Title: The Effect of a Musical Toy (Xylophone) on Pain, Fear, and Parental Satisfaction During Peripheral Intravenous Cannulation in Children Aged 3 to 6 Years
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Esra Nur Kocaaslan Mutlu (Other)
Responsible Party: Sponsor-Investigator, Esra Nur Kocaaslan Mutlu, Assistant Professor / Principal Investigator, Trakya University
Organization: Trakya University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TUTF-SBF-ENK-05
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Musical Toy (Xylophone) Group (Experimental): Children in this group will play with a colorful xylophone toy accompanied by a nurse before and during peripheral intravenous cannulation. The distraction is intended to reduce procedural pain and fear.
  Interventions: Behavioral: Musical Toy (Xylophone)
- Arm 2: Control Group (Other): Children in this group will undergo the standard IV insertion procedure with no distraction technique. Standard hospital protocol will be followed.
  Interventions: Other: Standard Care (in control arm)

INTERVENTIONS:
Behavioral: Musical Toy (Xylophone) — Children in this group will play with a colorful xylophone toy for 5 minutes before and during peripheral intravenous cannulation. A nurse (researcher) will assist the child in playing with the toy to distract them from the procedure. The toy will be cleaned between uses. This non-pharmacological method aims to reduce pain and fear.
  Arms: Arm 1: Musical Toy (Xylophone) Group
Other: Standard Care (in control arm) — Children in this group will receive routine peripheral intravenous cannulation according to standard hospital protocols. No distraction or behavioral intervention will be applied.
  Arms: Arm 2: Control Group

SUMMARY:
This randomized controlled trial investigates the effects of using a musical toy (xylophone) as a distraction technique during peripheral intravenous cannulation on pain, fear, and parental satisfaction in hospitalized children aged 3 to 6 years. The study will be conducted in the Pediatric Health and Diseases Clinic of Trakya University in Edirne, Turkey.

A total of 64 children will be randomly assigned to either the intervention group or the control group. Children in the intervention group will be encouraged to play with a xylophone, accompanied by a nurse, before and during the cannulation procedure. The control group will receive standard care without any distraction. Pain levels will be measured using the Wong-Baker FACES Pain Rating Scale, fear will be assessed using the Children's Fear Scale, and parental satisfaction will be evaluated using the PedsQL Healthcare Satisfaction Scale.

The primary objective is to evaluate whether the use of a musical toy during IV insertion reduces pain and fear in children. The secondary objective is to determine whether parental satisfaction with the healthcare experience is improved in the intervention group. Data will be collected before, during, and after the procedure.

This study is expected to contribute to the evidence base supporting the use of non-pharmacological methods in pediatric pain management and to promote child-friendly approaches in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 3 and 6 years
* Hospitalized and scheduled for peripheral intravenous cannulation
* No hearing or mental disabilities
* No chronic disease associated with pain
* No analgesic use in the past 6 hours
* One parent present during the procedure
* Both child and parent voluntarily agree to participate
* Intravenous cannulation to be performed in a single attempt
* Parent/guardian is literate

Exclusion Criteria:

* Children with hearing impairment or mental disabilities
* Use of analgesics within the last 6 hours
* Presence of chronic pain conditions
* Parental refusal to participate
* Failed intravenous cannulation attempt
* Illiterate parent/guardian
* Any parental mental disability
* Child or parent unwilling to participate

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
1. Pain Level | Within 5 minutes after the IV cannulation procedure
  Children's pain levels will be measured using the Wong-Baker FACES Pain Rating Scale, which ranges from 0 (no pain) to 5 (worst pain).
2. Fear Level | Before and within 5 minutes after the IV cannulation procedure
  Fear levels will be assessed using the Children's Fear Scale (CFS), which ranges from 0 (no fear) to 4 (extreme fear).

SECONDARY OUTCOMES:
Parental Satisfaction | Within 5-10 minutes after the procedure
  Parental satisfaction regarding their child's IV experience will be evaluated using the PedsQL Healthcare Satisfaction Scale. Scores range from 0 to 100, with higher scores indicating greater satisfaction.

IPD SHARING:
Plan to Share IPD: No